CLINICAL TRIAL: NCT01141842
Title: Prospective Clinical Study to Determine the Predictive Value of Sniffer Dogs to Identify Lung Cancer in the Exhalation of Patients With and Without Pulmonary Disease
Brief Title: Early Detection of Lung Tumors by Sniffer Dogs - Evaluation of Sensitivity and Specificity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Schillerhoehe Hospital (Other)
Responsible Party: Principal Investigator, Thorsten Walles, Principal Investigator, Schillerhoehe Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KSH-TCH-IIT-2010-1
Record Dates: First submitted 2010-05-11; First posted 2010-06-11 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Lung Cancer; Chronic Obstructive Airway Disease
Keywords: lung cancer; exhalation analysis; chronic obstructive pulmonary disease; cancer screening test
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- lung cancer (Experimental): breath samples of patients with confirmed lung cancer
  Interventions: Procedure: exhalation analysis of breath sample
- underlying lung disease (Active Comparator): patients with underlying lung disease and impairment in lung function
  Interventions: Procedure: exhalation analysis of breath sample
- healthy individual (Sham Comparator): healthy individual with no lung disease and no history of cancer including lung cancer
  Interventions: Procedure: exhalation analysis of breath sample

INTERVENTIONS:
Procedure: exhalation analysis of breath sample — breath sample is presented to sniffer dog in test tube
  Arms: lung cancer
Procedure: exhalation analysis of breath sample — breath sample is presented to sniffer dog in test tube
  Arms: underlying lung disease
Procedure: exhalation analysis of breath sample — breath sample is presented to sniffer dog in test tube
  Arms: healthy individual

SUMMARY:
Some groups reported that sniffer dogs can be applied to detect lung cancer in the exhaled breath of patients. Therefore, breath samples (BS) of patients are collected. Five sniffer dogs are trained to distinguish between the BS of patients with lung cancer and healthy individuals (controls). In a prospective, randomized blinded study the dog's ability to differentiate between BS of i) patients with lung cancer, ii) patients with inflammatory airway disease, but no evidence of cancer and iii) healthy individuals is tested.

DETAILED DESCRIPTION:
All breath samples (BS) are collected in patients on the basis of radiologic findings before any intervention (bronchoscopy, biopsy or surgery) has been performed. The allocation to study groups is made following diagnostic work up and surgery.

Three study groups are defined using the following inclusion and exclusion criteria:

* lung cancer: male & female, age 18-80, competent, confirmed lung cancer in diagnostic work up and surgery, no history or present other tumor disease
* healthy individual: male & female, age 18-80, competent, no history or present other tumor disease including lung cancer, no pathological lung function tests
* chronic obstructive lung disease: male & female, age 18-80, competent, no history or present other tumor disease including lung cancer, pathological lung function tests

For each patient, i) history, ii) present medication, iii) lung function tests are documented. For the lung cancer patients, the tumor stage following surgery is documented.

Five sniffer dogs are trained using BS of lung cancer patients and healthy individuals. After completion of the training the ability of the dogs to differentiate between the groups is tested:

* 5 BS are presented in 1 experiment:

  * Test I: lung cancer vs healthy individual
  * Test II: lung cancer vs chronic obstructive pulmonary disease
  * Test III: lung cancer vs healthy individuals & bronchitis
* for every experiment 1 BS of a lung cancer patient is used

  * the lung cancer sample is placed randomly in one of the five test tubes
  * the other test tubes are used for BS of healthy individuals or chronic obstructive pulmonary disease patients or both
  * neither the dog handler nor the dog know the loading of the test tubes
* experiments are repeated 5 to 10 times

For analysis, the sensitivity and specificity of the dog's reaction is determined.

The patient's medication, smoking habits, age and gender are analysed to rule out confounders or bias.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80
* competent
* confirmed lung cancer

Exclusion Criteria:

* history of other cancers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
presence of an heretofore unknown substrate in the exhalation sample of a patient with confirmed lung cancer | baseline
  number of individuals in the study cohort with confirmed lung cancer whose exhalation sample is correctly identified by sniffer dogs to contain an heretofore unknown substrate that is associated with lung cancer

SECONDARY OUTCOMES:
absence of an heretofore unknown substrate that is associated with lung cancer in patients with lung disease but excluded lung cancer | baseline
  number of individuals with confirmed impairment of lung function but exclusion of lung cancer whose exhalation sample is wrongly identified by sniffer dogs to contain a heretofore unknown substrate that is associated with lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Walles, MD, Principal Investigator — Schillerhoehe Hospital
Locations (2):
- Germany (2):
  - Schillerhoehe Hospital, Gerlingen
  - Praxis Heimann & Ehmann, Stuttgart

REFERENCES:
- [Background] Boedeker E, Friedel G, Walles T. Sniffer dogs as part of a bimodal bionic research approach to develop a lung cancer screening. Interact Cardiovasc Thorac Surg. 2012 May;14(5):511-5. doi: 10.1093/icvts/ivr070. Epub 2012 Feb 17. PMID 22345057
- [Result] Ehmann R, Boedeker E, Friedrich U, Sagert J, Dippon J, Friedel G, Walles T. Canine scent detection in the diagnosis of lung cancer: revisiting a puzzling phenomenon. Eur Respir J. 2012 Mar;39(3):669-76. doi: 10.1183/09031936.00051711. Epub 2011 Aug 18. PMID 21852337